CLINICAL TRIAL: NCT02658760
Title: Comparison of Dexmedetomidine and Bupivacaine With Bupivacaine Alone on the Quality of Ultrasonography Guided Fascia Iliaca Compartment Block in Adults Undergoing Femur Fracture Fixation Surgery
Brief Title: Dexmedetomidine and Bupivacaine With Bupivacaine in Ultrasonography Guided Fascia Iliaca Compartment Block in Adults
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamidreza Mahboobi (Other)
Responsible Party: Sponsor-Investigator, Hamidreza Mahboobi, Investigator, Hormozgan University of Medical Sciences
Organization: Hormozgan University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hums.Rec.1394.74
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Femoral Fractures
Keywords: Femoral Fractures
MeSH Terms: conditions — Femoral Fractures | interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bupivacaine (Experimental): 30cc of 0.25% bupivacaine
  Interventions: Drug: Bupivacaine
- Dexmedetomidine and bupivacaine (Active Comparator): 30cc of 0.25% bupivacaine and 2mg/kg dexmedetomidine
  Interventions: Drug: Dexmedetomidine; Drug: Bupivacaine

INTERVENTIONS:
Drug: Dexmedetomidine — dexmedetomidine plus placebo
  Arms: Dexmedetomidine and bupivacaine
Drug: Bupivacaine — dexmedetomidine and Bupivacaine

SUMMARY:
Few studies have reported the efficacy of adding dexmedetomidine to bupivacain for fascia illiaca compartment black. Comparison of dexmedetomidine and bupivacaine with bupivacaine alone on the quality of ultrasonography guided fascia iliaca compartment block in adults undergoing femur fracture fixation surgery at 2014.

ELIGIBILITY:
Inclusion Criteria:

* Adults with femural fracture

Exclusion Criteria:

* Hypersensitivity to drugs
* Neurological diseases
* Coagulation abnormalities
* Infection at the site of block

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Pain | 24 hours
  A point between 0 and 10 based on patient report

SECONDARY OUTCOMES:
Respiratory depression | 24 hours
  respiratory rate < 12/min
Hypotension | 24 hours
  Systolic blood pressure < 90 mmHg
Baradycardia | 24 hours
  Heart rate < 60/min

CONTACTS AND LOCATIONS:
Overall Officials: Nasim Abdi, Principal Investigator — Hormozgan University of Medical Sciences
Locations (1):
- Shahid Mohammadi hospital, Bandar Abbas, Hormozgan, Iran

IPD SHARING:
Plan to Share IPD: No